CLINICAL TRIAL: NCT00073944
Title: Phase I Pharmacology Study Of Oral And Intravenous BCX-1777 In Patients With Refractory T-Cell And Non-T-Cell Malignancies
Brief Title: BCX-1777 in Treating Patients With Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: BIOCRYST-1777BC-101; CDR0000341332 (Registry Identifier: PDQ (Physician Data Query)); CCF-5909
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2004-07

CONDITIONS: Cancer
Keywords: acute undifferentiated leukemia; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; atypical chronic myeloid leukemia, BCR-ABL1 negative; chronic eosinophilic leukemia; primary myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; essential thrombocythemia; intraocular lymphoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; polycythemia vera; previously treated myelodysplastic syndromes; primary central nervous system non-Hodgkin lymphoma; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; Waldenström macroglobulinemia; adenocarcinoma of the colon; adenocarcinoma of the esophagus; adenocarcinoma of the pancreas; adenocarcinoma of the rectum; recurrent adult brain tumor; recurrent adult primary liver cancer; recurrent colon cancer; recurrent esophageal cancer; recurrent gastric cancer; recurrent melanoma; recurrent ovarian epithelial cancer; recurrent pancreatic cancer; recurrent rectal cancer; adenocarcinoma of the stomach; adult anaplastic astrocytoma; adult glioblastoma; adult pilocytic astrocytoma; adult subependymoma; adenocarcinoma of the extrahepatic bile duct; recurrent extrahepatic bile duct cancer; recurrent cutaneous T-cell non-Hodgkin lymphoma; de novo myelodysplastic syndromes; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); adult diffuse astrocytoma; adult giant cell glioblastoma; adult gliosarcoma; T-cell large granular lymphocyte leukemia
MeSH Terms: conditions — Neoplasms; Leukemia, Biphenotypic, Acute; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Intraocular Lymphoma; Myeloproliferative Disorders; Polycythemia Vera; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia; Colonic Neoplasms; Adenocarcinoma Of Esophagus; Rectal Neoplasms; Brain Neoplasms; Carcinoma, Hepatocellular; Esophageal Neoplasms; Stomach Neoplasms; Melanoma; Carcinoma, Ovarian Epithelial; Pancreatic Neoplasms; Astrocytoma; Glioblastoma; Glioma, Subependymal; Bile Duct Neoplasms; Lymphoma, T-Cell, Cutaneous; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities; Gliosarcoma; Leukemia, Large Granular Lymphocytic

INTERVENTIONS:
Drug: forodesine hydrochloride

SUMMARY:
RATIONALE: BCX-1777 may stop the growth of cancer cells by blocking the enzymes necessary for their growth.

PURPOSE: Phase I trial to study the effectiveness of BCX-1777 in treating patients who have refractory cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of BCX-1777 in patients with refractory T-cell or non-T-cell malignancies.
* Determine the safety and dose-limiting toxicity of this drug in these patients.

Secondary

* Determine the pharmacokinetics of single oral and single and multiple IV doses of this drug in these patients.
* Determine the oral bioavailability of this drug in these patients.
* Determine, preliminarily, the antitumor activity of this drug in these patients.

OUTLINE: This is an open-label, nonrandomized, dose-escalation, multicenter study.

* Courses 1 and 2: Patients receive oral BCX-1777 on days 1 and 15* and BCX-1777 IV over 30 minutes on days 8* and 22*.
* Course 3: Beginning approximately 6 days* after the completion of courses 1 and 2, patients receive BCX-1777 IV over 30 minutes once daily on days 1-5 and 8-12 (total of 10 doses).

NOTE: *+/- 1 day

Patients with stable disease or better and no dose-limiting toxicity (DLT) may receive an additional 10-dose treatment course (as in course 3) after a 10- to 16-day drug-free interval.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BCX-1777 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT.

Patients are followed at 14 and 30 days.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Hematologic malignancy that is refractory to at least 1 prior curative treatment
  * Non-hematologic tumor that is refractory to at least 2 prior therapies, with or without measurable disease, including the following:

    * Gastrointestinal adenocarcinoma of 1 of the following sites:

      * Pancreatic
      * Biliary
      * Gastric
      * Colorectal
      * Esophageal
    * Melanoma
    * Ovarian cancer
    * Astrocytoma brain tumor
* Not immediately eligible for any other treatment that would be potentially curative or life-prolonging, in the opinion of the investigator

  * Patients who may be candidates for future bone marrow transplantation are eligible
* No brain metastases (other than astrocytomas)
* No clinically significant pleural effusion
* No complete tumor obstruction (e.g., bronchus, ureter, or bowel)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 50-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count greater than 50,000/mm^3
* Hematocrit stable without the need for transfusion (epoetin alfa support allowed)

Hepatic

* Bilirubin less than 1.5 times upper limit of normal (ULN) (unless due to Gilbert's syndrome)
* SGOT and SGPT less than 2 times ULN
* No active hepatitis B or C

Renal

* Creatinine clearance at least 50 mL/min

Cardiovascular

* No American Heart Association class III or IV cardiac disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No active systemic infection requiring IV antibiotics

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Concurrent corticosteroids allowed provided the patient is on a stable regimen

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Recovered from prior therapy

  * No grade 2-4 toxicity
* More than 3 weeks since prior antineoplastic and/or investigational therapy
* No other concurrent systemic antineoplastic or investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-04; Primary Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Shalaurov, MD, PhD, Study Chair — Inveresk Research Group, Incorporated
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States